CLINICAL TRIAL: NCT03522805
Title: Impact of Non-invasive Ventilation on Biomarkers in Hypercapnic COPD
Brief Title: Impact of Non-invasive Ventilation in Hypercapnic COPD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failure to accrue subjects. All activity has stopped & no analysis will be done on what has been collected.
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jeremy Orr, M.D., Assistant Clinical Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 161873
Record Dates: First submitted 2018-05-01; First posted 2018-05-11 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Copd; Chronic Obstructive Pulmonary Disease; Hypercapnia; Chronic Respiratory Failure; Hypoventilation
Keywords: copd; lung; non-invasive ventilation; hypercapnia; hypoventilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypercapnia; Hypoventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-invasive ventilation (Experimental): Subjects will undergo a baseline night with standard polysomnography, followed by a treatment night using non-invasive ventilation under polysomnography
  Interventions: Device: High-intensity non-invasive ventilation

INTERVENTIONS:
Device: High-intensity non-invasive ventilation — Single night of high-intensity non-invasive ventilation

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a highly prevalent condition worldwide and is a cause of substantial morbidity and mortality. Unfortunately, few therapies have been shown to improve survival. The importance of systemic effects and co-morbidities in COPD has garnered attention based on the observation that many patients with COPD die from causes other than respiratory failure, including a large proportion from cardiovascular causes. Recently, two high profile randomized trials have shown substantial improvements in morbidity and mortality with use of nocturnal non-invasive ventilation (NIV) in COPD patients with hypercapnia. Although the mechanisms by which NIV improves outcomes remain unclear, the important benefits of NIV might be cardiovascular via a number of mechanisms. In contrast to prior trials of NIV in COPD that did not show substantial benefit, a distinguishing feature of these encouraging recent NIV clinical trials was a prominent reduction of hypercapnia, which might be a maker or mediator of effective therapy. Alternatively, improvements might be best achieved by targeting a different physiological measure. Additional mechanistic data are therefore needed to inform future trials and achieve maximal benefit of NIV. Recent work in cardiovascular biomarkers has identified high-sensitivity troponin to have substantial ability to determine cardiovascular stress in a variety of conditions - even with only small changes. In COPD, a number of observational studies have shown that high-sensitivity troponin increases with worsening disease severity, and that levels increase overnight during sleep. This biomarker therefore presents a promising means to study causal pathways regarding the effect of NIV in patients with COPD. With this background, the investigator's overall goals are: 1) To determine whether the beneficial effect of non-invasive ventilation might be due to a reduction in cardiovascular stress, using established cardiovascular biomarkers, and 2) To define whether a reduction in PaCO2 (or alternative mechanism) is associated with such an effect.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with previously diagnosed severe COPD (FEV1 <50% predicted) and daytime hypercapnia (PaCO2 or TcCO2 > 45 mmHg)

Exclusion Criteria:

* Lung disease besides COPD (e.g., pulmonary fibrosis, bronchiectasis, pulmonary arterial hypertension) other than well controlled asthma
* Unrevascularized coronary artery disease, angina, prior heart attack or stroke, congestive heart failure
* Uncontrolled hypertension (SBP >160, DBP >95)
* Unwilling or unable to withhold CPAP during polysomnography
* Presence of tracheostomy
* Hospitalization within the past 90 days
* Prior peptic ulcer disease, esophageal varicies, or gastrointestinal bleeding (< 5 years)
* Prior gastric bypass surgery
* Anticoagulant use (other than aspirin) or bleeding diathesis (only for esophageal catheter placement)
* Chronic liver disease or end-stage kidney disease
* Allergy to any of the study medications
* Regular use of medications known to affect control of breathing (opioids, benzodiazepines, theophylline)
* Insomnia or circadian rhythm disorder
* Active illicit substance use or >3 oz nightly alcohol use
* Psychiatric disease, other than controlled depression
* Pregnancy
* Prisoners
* Cognitive impairment, unable to provide consent, or unable to carry out research procedures

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
Paired difference in morning level of high sensitivity troponin between baseline and NIV nights | 1 day
  Comparing morning levels of high sensitivity troponin between baseline and NIV nights

SECONDARY OUTCOMES:
Paired difference in overnight increase in high sensitivity troponin between baseline and NIV night | 1 day
  Troponin assay: Minimum 0, no maximum, with higher values worse.
Paired difference in sleep quality by Richards-Campbell Sleep Questionnaire between baseline and NIV night | 1 day
  Questionnaire: 5 questions, 0 to 100 on visual analog scale, with higher scores indicating better sleep. Total score reported as mean of 5 components.
Paired difference in sleep quality by arousal index between baseline and NIV night | 1 day
  Arousal index: Index reported as events/hour. Minimum 0, no maximum, with higher scores indicating worse sleep.
Paired difference in heart rate variability during sleep between baseline and NIV night | 1 day
  Comparing difference in heart rate variability during sleep between baseline and NIV night
Paired difference between Morning psychomotor vigilance testing score between baseline and NIV night | 1 day
  Psychomotor vigilance score: Reported as number of lapses. Minimum 0, no maximum, with higher values worse.
Paired difference in morning exhaled nitric oxide level between baseline and NIV night | 1 day
  Exhaled nitric oxide assay: Minimum 0, no maximumm with higher values worse.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy E Orr, MD, Principal Investigator — UCSD
Locations (1):
- University of California San Diego, San Diego, California, United States